CLINICAL TRIAL: NCT00538863
Title: Open-label Multi-center Safety Trial of Fentanyl Sublingual Spray (Fentanyl SL Spray) for the Treatment of Breakthrough Cancer Pain
Brief Title: Long-term Safety and Efficacy Study of Fentanyl Sublingual Spray for the Treatment of Breakthrough Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: INS-06-007; NCT00589004 (obsolete NCT alias)
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-08

CONDITIONS: Cancer; Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl sublingual spray titration (Experimental): Patients received fentanyl sublingual spray to treat up to a maximum of 4 breakthrough pain episodes per day with a minimum separation of 4 hours between treatments. Patients started at a dose of 100, 200, or 400 µg and titrated upward to a maximum dose of 1600 µg. Titration was stopped when the dose administered provided adequate analgesia for breakthrough pain without unacceptable side effects or the maximum titration period of 26 days was reached.
  Interventions: Drug: Fentanyl sublingual spray
- Fentanyl sublingual spray maintenance (Experimental): Patients received fentanyl sublingual spray up to a maximum of 4 times per day with a minimum separation of 4 hours between treatments for 90 days. Patients received a dose of 100 to 1600 µg determined in a previous study (INS-05-001, NCT00538850) or in the open-label dose titration period of the current study. The dose administered provided adequate analgesia for breakthrough pain without unacceptable side effects.
  Interventions: Drug: Fentanyl sublingual spray

INTERVENTIONS:
Drug: Fentanyl sublingual spray — Fentanyl sublingual spray in doses of 100, 200, 400, 600, 800, 1200, and 1600 µg

SUMMARY:
The purpose of this study was to assess the 90-day safety of fentanyl sublingual spray for the treatment of breakthrough cancer pain in subjects on around-the-clock opioids for their persistent cancer pain.

DETAILED DESCRIPTION:
This was an open-label multi-center study of the safety of fentanyl sublingual spray as a treatment for breakthrough cancer pain. The study medication was administered under the tongue as a simple spray and could be self-administered by patients or assisted by their caregivers. In addition to safety, there was a questionnaire to assess satisfaction with the study medication.

Subjects could enter this study by 1 of 2 routes:

* De novo subjects who meet the inclusion criteria and none of the exclusion criteria at the Screening Visit were enrolled into the Open-label Titration Period of the study. Upon successful completion of the titration period, patients entered the Open-label Maintenance Period.
* All patients who successfully completed the Double-blind Randomization Period and the Final Visit of study INS-05-001 (NCT00538850) were eligible to enter the Open-label Maintenance Period of this study.

ELIGIBILITY:
Inclusion Criteria:

All subjects who have completed the Double-blind Period and Final Visit of protocol INS-05-001(NCT00538850), Multicenter Randomized Double-blind Trial of Fentanyl Sublingual Spray for the Treatment of Breakthrough Cancer Pain are eligible for participation in this open-label extension study.

All de novo subjects must meet all of the following criteria to be eligible for participation in the study:

1. Male or female, > 18 years of age.
2. Diagnosis of cancer.
3. Opioid treatment. Patients who are treated with opioids are defined as those patients who are taking at least 60 mg of oral morphine/day, at least 25 µg of transdermal fentanyl/hour, at least 30 mg of oxycodone/day, at least 8 mg of oral hydromorphone/day or an equianalgesic dose of another opioid for > 7 days for cancer-related pain.
4. Experience persistent pain related to the cancer or its treatment of moderate or lesser intensity in the 24 hours prior to assessment by a verbal rating scale at the Screening Visit.
5. Experience on average 1 to 4 breakthrough cancer pain episodes per day usually at least partially controlled by supplemental medication of at least 5 mg immediate-release morphine or an equivalent short-acting opioid (eg, oxycodone, hydrocodone, or codeine with acetaminophen).
6. Able to evaluate pain relief, assess medication performance, report adverse events (AEs), report use of the study drug or supplemental medication (a caregiver may provide the subject the medication).
7. Able and willing to give informed consent.
8. Women of childbearing potential must have a) a negative urine pregnancy test, b) not be breast feeding and c) agree to practice a reliable form of contraception.

Exclusion Criteria:

1. Intolerable side effects to opioids or fentanyl.
2. Rapidly increasing/uncontrolled pain.
3. A history of major organ system impairment or disease, that in the Investigator's or his/her designee's opinion could increase the risk associated with the use of opioids.
4. Uncontrolled hypertension (systolic blood pressure [BP] > 180 mm Hg or diastolic BP > 90 mm Hg on 2 occasions at least 6 hours apart) despite antihypertensive therapy, or has a history of hypertensive crisis within the past 2 years.
5. A recent history (within the past 2 years) of transient ischemic attacks, neural vascular disease, stroke, or cerebral aneurysms.
6. Serum creatinine, ALT or AST that is greater than 3 times the upper limit of normal.
7. Diagnosis of sleep apnea.
8. Brain metastases with signs or symptoms of increased intracranial pressure.
9. Inability to assess pain or response to pain medications for any reason, including psychiatric disorder, concurrent medical disorder, or concomitant therapy.
10. Has used methadone within 14 days of the Screening Visit.
11. Received an investigational study product(s) within 30 days of the Screening Visit.
12. Use of monoamine oxidase (MAO) inhibitors within 14 days of the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2007-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Dillaha, MD, Study Director — Chief Medical Officer, Insys Therapeutics Inc
Locations (52):
- United States (40):
  - Huntsville, Alabama
  - Winfield, Alabama
  - Glendale, Arizona
  - Scottsdale, Arizona
  - Laguna Hills, California
  - Loma Linda, California
  - Los Gatos, California
  - San Mateo, California
  - Bradenton, Florida
  - Lake Worth, Florida
  - Miami, Florida
  - Winter Park, Florida
  - Newnan, Georgia
  - Chicago, Illinois
  - Skokie, Illinois
  - Zion, Illinois
  - Elkhart, Indiana
  - Bethesda, Maryland
  - Southfield, Michigan
  - Edina, Minnesota
  - Jefferson City, Missouri
  - Great Falls, Montana
  - Kalispell, Montana
  - Missoula, Montana
  - Voorhees Township, New Jersey
  - Flat Rock, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Dayton, Ohio
  - Eugene, Oregon
  - Altoona, Pennsylvania
  - Danville, Pennsylvania
  - Lemoyne, Pennsylvania
  - Kingsport, Tennessee
  - Bellaire, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Port Sam Houston, Texas
  - Tacoma, Washington
  - Appleton, Wisconsin
- Canada (4):
  - Oakville, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- India (8):
  - Ahmedabad, India
  - Bangalore, India
  - Bhopal, India
  - Hyderabad, India
  - Jaipur, India
  - Mumbai, India
  - Nashik, India
  - Pune, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of patients in the fentanyl sublingual spray maintenance group includes 179 patients who completed the fentanyl sublingual spray titration period of the study plus 90 patients who entered the study directly in the maintenance period.
Pre-assignment Details: Five patients who completed the titration period did not start the maintenance period due to failure to determine a dose in the titration period (n=1), withdrawal from the study (n=3), and adverse event (n=1).
Groups:
- Fentanyl Sublingual Spray: In the titration period, patients were titrated upward to a maximum dose of 1600 µg fentanyl sublingual spray. In the maintenance period, patients received a dose of 100 to 1600 µg fentanyl sublingual spray determined in a previous study (INS-05-001, NCT00538850) or in the titration period of the current study.
Period: Open-label Titration
Arm/Group | Fentanyl Sublingual Spray
Started | 229
Completed | 184
Not Completed | 45
Period: Open-label Maintenance
Arm/Group | Fentanyl Sublingual Spray
Started | 269 (Five participants who completed the titration period did not start the maintenance period.)
Completed | 163
Not Completed | 106

BASELINE CHARACTERISTICS:
Population: The total number of patients enrolled in the study is 319.
Arm/Group | Fentanyl Sublingual Spray
Number analyzed (Participants) | 319
Age Continuous [Mean (Standard Deviation); unit: years]
  Titration Period | 54.1 (12.5)
  Maintenance Period | 53.6 (12.2)
Sex/Gender, Customized [Number; unit: Participants]
  Titration period - Female | 117
  Titration period - Male | 112
  Maintenance period - Female | 141
  Maintenance period - Male | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Experienced 1 or More Adverse Events
Time Frame: Baseline to end of the study (up to 116 days)
Population: Safety population: All patients who received study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | Fentanyl Sublingual Spray Titration | Fentanyl Sublingual Spray Maintenance
Number analyzed (Participants) | 229 | 269
Percentage of patients | 59.0 | 80.7

ADVERSE EVENTS:
Time Frame: All adverse events were followed to resolution, an outcome had been reached, stabilization, or the event was otherwise explained regardless of whether the subject was still participating in the study (up to 150 days).
Description: Safety population: All patients (n=319) who received study medication. The number of patients in the fentanyl sublingual spray maintenance group includes 179 patients who completed the fentanyl sublingual spray titration period of the study plus 90 patients who entered the study directly in the maintenance period.
Arm/Group | Fentanyl Sublingual Spray Titration | Fentanyl Sublingual Spray Maintenance
Serious Adverse Events (participants affected / at risk) | 33/229 | 178/269
Other Adverse Events (participants affected / at risk) | 194/229 | 269/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Sublingual Spray Titration (N=229) | Fentanyl Sublingual Spray Maintenance (N=269)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Disease progression (General disorders) | 2 | 5
Bacterial sepsis (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Sepsis syndrome (Infections and infestations) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 60
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Lobar pneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Real failure acute (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Sublingual Spray Titration (N=229) | Fentanyl Sublingual Spray Maintenance (N=269)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 65
Vomiting (Gastrointestinal disorders) | 27 | 43
Nausea (Gastrointestinal disorders) | 30 | 28
Somnolence (Nervous system disorders) | 23 | 10
Oedema peripheral (General disorders) | 7 | 31
Constipation (Gastrointestinal disorders) | 13 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 28
Asthenia (General disorders) | 4 | 26
Fatigue (General disorders) | 7 | 23
Application site irritation (General disorders) | 17 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 20
Dizziness (Nervous system disorders) | 16 | 3
Pyrexia (General disorders) | 11 | 18
Anaemia (Blood and lymphatic system disorders) | 3 | 17
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 17
Anxiety (Psychiatric disorders) | 3 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 15
Anorexia (Metabolism and nutrition disorders) | 2 | 14
Dehydration (Metabolism and nutrition disorders) | 1 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No